CLINICAL TRIAL: NCT02761096
Title: Effect of Acupuncture on Inflammation and Immune Function After Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Kyunghee University (Other)
Responsible Party: Principal Investigator, Seong-Uk Park, KMD, PhD, Kyunghee University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20152152
Record Dates: First submitted 2016-04-27; First posted 2016-05-04 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Unruptured Cerebral Aneurysm; Hemifacial Spasm; Brain Tumor
MeSH Terms: conditions — Hemifacial Spasm; Brain Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Experimental): The acupuncture intervention will start no more than 48 hours after craniotomy and will be given once a day for 6 days (a total of 6 sessions within 8 days). It will be given in addition to conventional treatments. All interventions will be performed by one Korean Medicine doctor with over 5 years of working experience with a college education of 6 years. This doctor will be trained in the study protocol before the start of the trial.
  Interventions: Device: acupuncture; Other: conventional treatment
- Control group (Other): The subjects in the control group will only receive conventional treatment. This involves general management after craniotomy in the department of neurosurgery.
  Interventions: Other: conventional treatment

INTERVENTIONS:
Device: acupuncture — Acupuncture, electroacupuncture, and intradermal acupuncture will be performed at every session.
  Sterile disposable stainless steel acupuncture needles (0.25 mm × 30 mm) will be used. Acupuncture needles will be inserted bilaterally at the following acupuncture points: LI4, LI11, PC6, ST36, GB39 and LR3, and GV20. If GV20 is close to the surgical site, this acupoint may be excluded.
  An electric stimulator will be connected to the handle of each needle at LI4, LI11, ST36, and LR3 and a current of 5 Hz will be applied.
  After the needles are removed, intradermal acupuncture needles with tape (DB130A; 0.25 mm × 1.5mm) will be inserted at the same acupoints (LI4, LI11, PC6, ST36, GB39, and LR3 bilaterally, and GV20) and left in place until the next session.
  Arms: Study group
Other: conventional treatment — The subjects in the control group will only receive conventional treatment. This involves general management after craniotomy in the department of neurosurgery and includes stabilizing vital signs, pain control, prevention and treatment of infections, and other IV fluid or drug therapy required based on the condition of the patient.

SUMMARY:
The aim of this study is to evaluate the effect of acupuncture on inflammation and immune function after craniotomy. This study will be a single-center, parallel group clinical trial that will be conducted at Kyung Hee University Hospital at Gangdong, Seoul, Korea.

DETAILED DESCRIPTION:
For Study group, The intervention will start no more than 48 hours after craniotomy and will be given once a day for 6 days (a total of 6 sessions within 8 days). Acupuncture, electroacupuncture, and intradermal acupuncture will be performed at every session.

For Control group, The subjects in the control group will only receive conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria in order to be included:

1. planning to undergo regular craniotomy performed for an unruptured aneurysm, facial spasm, or brain tumor;
2. age > 18 years;
3. acupuncture treatment that can start within 48 h after craniotomy;
4. voluntary participation and provision of signed informed consent form.

Exclusion Criteria:

Participants with any of the following conditions will be excluded:

1. serum C-reactive protein (CRP) level ≥ 1.0 mg/dl before craniotomy;
2. a condition other than an unruptured aneurysm, facial spasm, or brain tumor as an indication for craniotomy;
3. craniotomy performed for infectious brain diseases such as brain abscess or subdural empyema;
4. medication use that can affect the immune system or white blood cell (WBC) count, such as immunosuppressive drugs, steroids, or anticancer drugs or use of these medications within one month prior to the craniotomy;
5. a history of surgery at the same site;
6. emergency surgery; or
7. a severe medical disease, e.g. congestive heart failure, chronic renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-04; Primary Completion 2017-05 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Serum CRP | 2 days after surgery
  Turbidimetric immunoassay will be performed for measurement of CRP. A blood sample will be drawn from the brachial vein at a fixed time in the morning before breakfast.

SECONDARY OUTCOMES:
Serum CRP | within 48 h before the surgery, 4 days after surgery and 7 days after surgery
  Turbidimetric immunoassay will be performed for measurement of CRP. A blood sample will be drawn from the brachial vein at a fixed time in the morning before breakfast.
Serum erythrocyte sedimentation rate (ESR) | within 48 h before the surgery, 2 days after surgery, 4 days after surgery and 7 days after surgery
  The photometrical capillary method will be performed for measurement of ESR. A blood sample will be drawn from the brachial vein at a fixed time in the morning before breakfast.
Serum TNF-α | within 48 h before the surgery, 2 days after surgery, 4 days after surgery and 7 days after surgery
  Enzyme-linked immunosorbent assay (ELISA) will be performed for measurement A blood sample will be drawn from the brachial vein at a fixed time in the morning before breakfast.
Serum IL-1β | within 48 h before the surgery, 2 days after surgery, 4 days after surgery and 7 days after surgery
  Enzyme-linked immunosorbent assay (ELISA) will be performed for measurement A blood sample will be drawn from the brachial vein at a fixed time in the morning before breakfast.
Serum IL-6 | within 48 h before the surgery, 2 days after surgery, 4 days after surgery and 7 days after surgery
  Enzyme-linked immunosorbent assay (ELISA) will be performed for measurement A blood sample will be drawn from the brachial vein at a fixed time in the morning before breakfast.
fever | During the post operation day to 7 days after operation day. Body temperature will be measured at 6:00, 10:00, 18:00, and 22:00 every day.
  Any fever with a body temperature over 38℃ will be recorded on the case report form.
use of additional antibiotics | During the post operation day to 7 days after operation day
  Use of additional antibiotics will be recorded on the case report form.
infection sign | During the post operation day to 7 days after operation day,
  Infections such as pneumonia or urinary tract infections will be recorded on the case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Uk Park, KMD, PhD, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho SY, Yang SB, Shin HS, Lee SH, Koh JS, Kwon S, Jung WS, Moon SK, Park JM, Ko CN, Park SU. Anti-inflammatory and immune regulatory effects of acupuncture after craniotomy: study protocol for a parallel-group randomized controlled trial. Trials. 2017 Jan 10;18(1):10. doi: 10.1186/s13063-016-1712-7. PMID 28069040